CLINICAL TRIAL: NCT04682639
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Etrasimod in Adult Subjects With Eosinophilic Esophagitis
Brief Title: A Study to Assess the Safety and Efficacy of Oral Etrasimod in Adult Participants With Eosinophilic Esophagitis
Acronym: VOYAGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: APD334-206; C5041009 (Other: Alias Study Number); 2020-003226-23 (EudraCT Number)
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic esophagitis; Esophageal eosinophilia; Etrasimod; APD334; EoE; Eosinophilic oesophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Etrasimod Dose 1 (Experimental)
  Interventions: Drug: Etrasimod
- Etrasimod Dose 2 (Experimental)
  Interventions: Drug: Etrasimod
- Placebo and Etrasimod (Placebo Comparator): Participants will receive etrasimod matching placebo tablet during the Double-Blind Treatment Period and etrasimod tablet during the Extension Treatment Period.
  Interventions: Drug: Placebo; Drug: Etrasimod

INTERVENTIONS:
Drug: Etrasimod — Participants will receive etrasimod tablet by mouth, once daily during the 24-week Double-Blind and 28-week Extension Treatment Periods.
  Other Names: APD334
  Arms: Etrasimod Dose 1; Etrasimod Dose 2
Drug: Placebo — Participants will receive etrasimod matching placebo tablet by mouth, once daily during the 24-week Double-Blind Treatment Period.
  Arms: Placebo and Etrasimod
Drug: Etrasimod — Participants will receive etrasimod tablet by mouth, once daily during the 28-week Extension Treatment Period.
  Other Names: APD334
  Arms: Placebo and Etrasimod

SUMMARY:
The purpose of this study is to determine whether oral etrasimod is a safe and effective treatment for active eosinophilic esophagitis (EoE) in adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Have an eosinophilic esophagitis (EoE) diagnosis prior to screening and histologically active disease with an esophageal peak eosinophil count (PEC) of ≥ 15 eosinophils per high powered field (eos/hpf)
* Have dysphagia, defined as solid food going down slowly or getting stuck in the throat with an average frequency of ≥ 2 episodes per week over 2 weeks during the Screening period

Inclusion Criteria for the Extension Treatment Period

* Completion of the Week 24 study visit [including esophagogastroduodenoscopy (EGD)]
* Compliance with study procedures during the Double-Blind Treatment Period as assessed by the Investigator
* No notable safety concerns during the Double-Blind Treatment Period, as determined by the Investigator
* Willing to comply with all study visits and procedures for the Extension Treatment Period

Exclusion Criteria:

* History of any of the non-EoE conditions or procedures that may interfere with the evaluation of or affect the histologic (eg eosinophilic gastritis), endoscopic (eg, high-grade esophageal stenosis), or symptom endpoints (eg, esophageal resection) of the study
* Undergone dilation of an esophageal stricture within 12 weeks prior to Screening EGD
* Use of corticosteroids for the treatment of EoE within 8 weeks prior to Screening EGD
* Discontinue, initiate, or change dosing (dosage/frequency) of the following therapies for EoE within 8 weeks prior to Screening EGD. Participants on any of the following therapy need to stay on a stable regimen during study participation:

  1. Elemental diet
  2. EoE food trigger elimination diet
  3. Proton pump inhibitor (PPI) therapy
* Used any immunotherapy/desensitization including oral immunotherapy (OIT) or sublingual immunotherapy (SLIT) within 12 months prior to the Screening EGD. Note: Stable (ie, ≥ 6 months prior to the Screening EGD) subcutaneous immunotherapy (SCIT) is permitted. Participants on SCIT need to stay on a stable treatment during study participation
* Used any protocol-specified immunomodulatory therapies within the protocol-specified timeframe prior to Baseline (eg, dupilumab, benralizumab, omalizumab, or infliximab within 12 weeks; a sphingosine-1-phosphate receptor modulator at any time)
* Use of any investigational agent or device within 12 weeks prior to Baseline
* Females who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (253):
- United States (218):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - GastroHealth - St. Vincent's East, Birmingham, Alabama
  - Digestive Health Specialists, Dothan, Alabama
  - Dothan Eyecare - Dr. Brent McKinley (OCT Procedure Only), Dothan, Alabama
  - Dothan Surgery Center (Colonoscopy Location), Dothan, Alabama
  - Pulmonary Associates (PFT Procedure Only, Second Location ), Dothan, Alabama
  - Flowers Hospital (PFT Procedure Only), Dothan, Alabama
  - Avant Research Associates, LLC, Huntsville, Alabama
  - Crestwood Medical Center, Huntsville, Alabama
  - Baily Cove Eye Care, Huntsville, Alabama
  - Madison Surgery Center, Madison, Alabama
  - Alabama Eye MD, Vestavia Hills, Alabama
  - Arizona Retina Institute/ Phoenix Retina Associates(OCT), Peoria, Arizona
  - SimonMed Imaging (Imaging), Peoria, Arizona
  - Arizona Digestive Health - Sun City, Sun City, Arizona
  - Sun City Endoscopy Center (Endoscopy), Sun City, Arizona
  - Little Rock Eye Clinic, Little Rock, Arkansas
  - Four Seasons Allergy and Asthma, Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Premier Gastroenterology Endoscopy Center, Little Rock, Arkansas
  - Premier Gastroenterology, Little Rock, Arkansas
  - Isight Vision Care, Fountain Valley, California
  - Mile Square Surgery Center, Fountain Valley, California
  - Pulmonary & Sleep Consultants, Fountain Valley, California
  - Paragon Rx Clinical, Inc., Garden Grove, California
  - Inland Pulmonary Specialists [PFT Only], Lake Elsinore, California
  - Advanced Endoscopy and Pain Center - EGD & Biopsy Collection, Lancaster, California
  - Advanced Endoscopy and Pain Center, Lancaster, California
  - Antelope Valley Eye Care - OCT, Lancaster, California
  - Antelope Valley Eye Care, Lancaster, California
  - Antelope Valley Lung and Sleep Institute, Lancaster, California
  - Apollo Surgery Center, Lancaster, California
  - AV Pediatrics, Allergy and Family Medicine - PFT, Physical Exams, Lab Reviews, ECG Reviews, Lancaster, California
  - Gastro Care Institute, Lancaster, California
  - Jatinder S. Pruthi, MD FACG CPI - Physical Exams, Lab Reviews, ECG Reviews, Lancaster, California
  - Om Research LLC, Lancaster, California
  - Clinical Trials Unit, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - USC IDS Pharmacy, Los Angeles, California
  - Advanced Vision Care (OCT), Los Angeles, California
  - United Surgery Center Murrieta [Endoscopy Only], Murrieta, California
  - United Medical Doctors, Murrieta, California
  - California Eye Professionals [OCT Only], Temecula, California
  - United Surgery Center Temecula [Endoscopy Only], Temecula, California
  - RecioMed Clinical Research Network, Inc, Boynton Beach, Florida
  - Steelgate, Bradenton, Florida
  - Bay Area Chest Physicians, P.A., - Pulmonary Function Test, Clearwater, Florida
  - West Coast Endoscopy Center, Clearwater, Florida
  - West Coast Endoscopy, Clearwater, Florida
  - MACULA CENTER Dana M. Deupree, M.D., F.A.C.S (OCT), Clearwater, Florida
  - Northwood Vision Optical Coherence Tomography (OCT), Clearwater, Florida
  - Safety Harbor Surgery Center, Clearwater, Florida
  - Gastro Florida (Regulatory & Administrative Duties), Clearwater, Florida
  - Beraja Medical Institute (OCT), Coral Gables, Florida
  - Bayfront Health Seven Rivers (Liver Biopsy Location), Crystal River, Florida
  - Citrus Surgery and Endoscopy Center (EGD Location), Crystal River, Florida
  - Advanced Eye Center, Hialeah, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - West Coast Eye Institute (OCT Procedure Only), Inverness, Florida
  - Suncoast Endoscopy Center (EGD Location), Inverness, Florida
  - Jupiter Outpatient Surgery Center, Jupiter, Florida
  - Central Florida Sleep Diagnostic & Treatment Center, Lakeland, Florida
  - Auzmer Research, Lakeland, Florida
  - West Coast Eye Institute (OCT Procedure Only), Lecanto, Florida
  - The Endoscopy Center (Endoscopy Procedure), Miami, Florida
  - Research Associates of South Florida, Miami, Florida
  - Juan Barrio, MD (PFT when needed), Miami, Florida
  - Florida Eye Specialists and Cataract Institute, Riverview, Florida
  - Dr. Dennis Bassetti, MD, Sebring, Florida
  - Highlands Eye Institute, P.A., Sebring, Florida
  - The Surgery and Endoscopy Center, Sebring, Florida
  - Ambulatory Surgery Center, Tampa, Florida
  - Pulmonology & Sleep Disorders, Tampa, Florida
  - Day Surgery Center, Winter Haven, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Peachtree Allergy and Asthma Clinica - Pulmonary Function Test, Atlanta, Georgia
  - Piedmont Hospital- DLCO, Atlanta, Georgia
  - Ross Eyecare - Opthalmoscopy and OCT, Atlanta, Georgia
  - Georgia Eye Partners, Decatur, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Atlanta Endoscopy Center LTD, Decatur, Georgia
  - Pulmonary & Sleep Specialist, Decatur, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Grand Teton Surgical Center, Idaho Falls, Idaho
  - Idaho Falls Pulmonary/ Sleep and Critical Care Specialists (PFT procedure only), Idaho Falls, Idaho
  - Premier Eye Care of Eastern Idaho (OCT procedure only), Idaho Falls, Idaho
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Glen Endoscopy Center (Endoscopy Facility), Glenview, Illinois
  - GI Alliance (PFT), Gurnee, Illinois
  - Illinois Gastroenterology Group-Gurnee (Patients Seen; IP Delivered), Gurnee, Illinois
  - Medical Eye Services LTD (Ophthalmoscopy with OCT), Gurnee, Illinois
  - North Shore Endoscopy Center (Endoscopy), Lake Bluff, Illinois
  - Libertyville Imaging Center (Diagnostic Imaging), Libertyville, Illinois
  - Clark Memorial Health (PFTs), Jeffersonville, Indiana
  - One Anesthesia, AACC Division, Jeffersonville, Indiana
  - Baptist Health Floyd (PFTs), New Albany, Indiana
  - Gastroenterology Health Partners, PLLC, (IP), New Albany, Indiana
  - John Kenyon Eye Center (OCT), New Albany, Indiana
  - One Anesthesia, PLLC, New Albany, Indiana
  - Physicians Medical Center (Endoscopies), New Albany, Indiana
  - Quest, Lenexa, Kansas
  - Cotton O'Neil Clinic (OCT Procedure Only), Topeka, Kansas
  - Cotton O'Neil Clinic (PFT Procedure Only), Topeka, Kansas
  - Cotton O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Acadiana Endoscopy Center, Inc, Lafayette, Louisiana
  - Acadiana Gastroenterology Associates, Lafayette, Louisiana
  - Combined Gastro Research, LLC, Lafayette, Louisiana
  - Gastroenterology Clinic of Acadiana (IP address), Lafayette, Louisiana
  - Lafayette General Endoscopy Center, Lafayette, Louisiana
  - Lafayette Family Eye Care, Lafayette, Louisiana
  - M Health Fairview Clinics and Surgery Center, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Minnesota Health Clinical research unit, Minneapolis, Minnesota
  - University of Minnesota Health Opthalmology Clinic, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Celerion, Inc., Lincoln, Nebraska
  - Del Negro & Senft Eye Associates, Brick, New Jersey
  - Allied Health Clinical Research Organization, LLC (IP Address), Brick, New Jersey
  - Seashore Surgical Institute, Brick, New Jersey
  - Shore Pulmonary, PA, Brick, New Jersey
  - Allied Health Clinical Research Organization, LLC, Freehold, New Jersey
  - Del Negro & Senft Eye associates, Neptune City, New Jersey
  - Del Negro & Senft eye Associates, Red Bank, New Jersey
  - lnvestigational Drug Services, University of North Carolina Hospitals (IP storage address), Chapel Hill, North Carolina
  - UNC Clinical Research Eastowne, Chapel Hill, North Carolina
  - UNC Hospitals Pulmonary Function Lab (PFT and DLCO procedures only), Chapel Hill, North Carolina
  - University of North Carolina - Memorial Hospital, Chapel Hill, North Carolina
  - UNC Endoscopy Center at Meadowmont, Chapel Hill, North Carolina
  - UNC Hospitals Pulmonary Specialty Clinic (PFT and DLCO procedures only), Chapel Hill, North Carolina
  - UNC Kittner Eye Center (OCT procedure only), Chapel Hill, North Carolina
  - Clinical and Translational Research Center Outpatient Unit, Chapel Hill, North Carolina
  - Duke Medical Plaza North Duke Street, Durham, North Carolina
  - Duke Eye Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Investigational Drug Services (Pharmacy), Durham, North Carolina
  - Coastal Research Institute, Fayetteville, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - UNC Gastroenterology at Hillsborough, Hillsborough, North Carolina
  - Brier Creek Medical Pavilion, Raleigh, North Carolina
  - Geauga Sleep Center (PFT Only), Chardon, Ohio
  - Leon A. Reid, III, M.D. (OCT), Cincinnati, Ohio
  - Cincinnati Eye Institute (ophthalmic and OCT exams), Cincinnati, Ohio
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Gastro Health Research, Cincinnati, Ohio
  - Ohio GI and Liver Institute, Cincinnati, Ohio
  - Tristate Endoscopy Center (Endoscopy), Cincinnati, Ohio
  - UC Health Hoxworth (ophthalmic and OCT only), Cincinnati, Ohio
  - UC Health Physicians Office Clifton (where subjects seen), Cincinnati, Ohio
  - UC Health Pulmonary (PFT Location), Cincinnati, Ohio
  - University of Cincinnati Medical Center Diagnostic Center (Endoscopy location), Cincinnati, Ohio
  - UC Health Pulmonary (Pulmonary Function Testing), Cincinnati, Ohio
  - New Horizons Clinical Research (PFT), Cincinnati, Ohio
  - University Endoscopy Center (Endoscopy location), Cincinnati, Ohio
  - UC Health/Division of Digestive Diseases (where subjects seen), Cincinnati, Ohio
  - Erdey Searcy Eye Group, Columbus, Ohio
  - Ohio Gastroenterology Group, Dublin, Ohio
  - Great Lakes Medical Research, LLC, Mentor, Ohio
  - The Endoscopy Center of Lake County, Mentor, Ohio
  - Vitreo Retinal Consultants (OCT only), Painesville, Ohio
  - Lake Pulmonary Associates (PFT only), Willoughby, Ohio
  - Retina Specialists of Ohio(OCT only), Willoughby Hills, Ohio
  - Norman Endoscopy Center, Norman, Oklahoma
  - Digestive Disease Specialists, Inc. Endoscopy Lab, Oklahoma City, Oklahoma
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Pulmonary Physicians of Oklahoma, Oklahoma City, Oklahoma
  - Retinal Center of Oklahoma, Oklahoma City, Oklahoma
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Johnston Eye, Oklahoma City, Oklahoma
  - West Shore Endoscopy Center, Camp Hill, Pennsylvania
  - Medical Arts Allergy,PC (PFT Only), Harrisburg, Pennsylvania
  - Farrel Opthalmology(OCT only), Harrisburg, Pennsylvania
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - Harrisburg Eye Associates (OCT only), Harrisburg, Pennsylvania
  - Penn State Health Medical Group - Lemoyne (PFT only), Lemoyne, Pennsylvania
  - Investigational Drug Services, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Tower Health Reading Hospital, West Reading, Pennsylvania
  - Berks Center for Digestive Health, Wyomissing, Pennsylvania
  - Berks Schuylkill Respiratory Specialists "PFT Procedure Only", Wyomissing, Pennsylvania
  - Eye Consultants of Pennsylvania, PC "OCT Procedure Only", Wyomissing, Pennsylvania
  - Regional Gastroenterology Associates of Lancaster, Ltd., Wyomissing, Pennsylvania
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - Franklin Woods Community Hospital (PFT Only), Johnson City, Tennessee
  - Pulmonary Associates of ET/Jeff Farrow, MD - PFT only, Johnson City, Tennessee
  - The Regional Eye Center - OCT only, Kingsport, Tennessee
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - Vanderbilt GI Endoscopy Lab at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University Medical Center - GI Research Office, Nashville, Tennessee
  - Vanderbilt University Medical Center GI Endoscopy Lab, Nashville, Tennessee
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Vanderbilt Pulmonary Medicine, Nashville, Tennessee
  - Vanderbilt University Medical Center - Digestive Disease Center, Nashville, Tennessee
  - Vanderbilt University Medical Center - Heart Station, Nashville, Tennessee
  - Digestive Health Center (Endoscopy), Dallas, Texas
  - Precision for Medicine, Houston, Texas
  - CHRJSTUS Santa Rosa Physicians Ambulatory Surgery Center-new Braunfels(Endoscopy), New Braunfels, Texas
  - Tyrus Schroeder (PFT), New Braunfels, Texas
  - The Eye Place Jenny Fan, OD (OCT Only), Plano, Texas
  - Pulmonary Medicine Consultants (PFT with DCLO only), Richardson, Texas
  - Advanced Imaging, San Marcos, Texas
  - Central Texas Eye Center (OCT), San Marcos, Texas
  - CHRJSTUS Santa Rosa Physicians Ambulatory Surgery Center - San Marcos (Endoscopy), San Marcos, Texas
  - Bay Area Houston Endoscopy Center (Endoscopy), Webster, Texas
  - Coastal Eye Associates (OCT), Webster, Texas
  - GI Alliance (Patients Seen), Webster, Texas
  - Houston Lung and Sleep Clinic, PA (PFT), Webster, Texas
  - University of Utah Gastroenterology Division Research, Salt Lake City, Utah
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - University Of Utah School Of Medicine, Salt Lake City, Utah
  - Chesapeake Pulmonary and Critical Care Medicine (PFT Only), Chesapeake, Virginia
  - Gastroenterology Associates of Tidewater - Endoscopy Center, Chesapeake, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Harman Eye Center (OCT only), Forest, Virginia
  - Lynchburg Pulmonary Associates, Inc. (PFT only), Lynchburg, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Wagner Macula and Retina Center (OCT only), Norfolk, Virginia
  - Sleep Specialists of Tidewater - Virginia Beach (PFT Only), Virginia Beach, Virginia
- Australia (23):
  - Sunshine University Private Hospital, Birtinya, Queensland
  - Mater Misericordiae Ltd, Brisbane South, Queensland
  - Buderim Eye Centre (OCT Facility), Buderim, Queensland
  - Dr Shiran DeSilva Respiratory Clinic, Mackay, Queensland
  - Mackay Discount Drug Store, Mackay, Queensland
  - Mater Misericordiae Hospital, Mackay, Queensland
  - Queensland X-Ray, Mackay, Queensland
  - Vision Eye Institute Mackay, Mackay, Queensland
  - Coastal Digestive Health, Maroochydore, Queensland
  - Coral Sea Clinical Research Institute, North Mackay, Queensland
  - Elizabeth Specialist Suites (PFT Facility), Elizabeth Vale, South Australia
  - Lyell McEwin Hospital., Elizabeth Vale, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Modbury Hospital (OCT Facility), Modbury, South Australia
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Eastern Health, Box Hill, Victoria
  - Box Hill Eye Surgeons (OCT Facility), Box Hill North, Victoria
  - Retina Specialists Victoria (OCT Facility), Camberwell, Victoria
  - The Northern Hospital, Epping, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Vision Eye Institute, Melbourne, Victoria
  - MCES Practice Pty Ltd operating as Comprehensive Eye Surgeons (OCT Facility), Bellfield
  - Queensland Respiratory Services ,Pulse Oceanside Medical{PFT Facility ), Birtinya
- Belgium (3):
  - AZ St Lucas Brugge, Bruges
  - AZ Delta, Roeselare
  - Centre Hospitalier Wallonie Picarde (CHWAPI), Tournai
- Mount Sinai Services Inc. Dr George Charames, Toronto, Ontario, Canada
- Precision for Medicine GmbH, Berlin, Germany
- Amsterdam UMC, location AMC, Amsterdam, Netherlands
- Spain (3):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - University Hospital Zurich, Zurich
  - Universitätsspital Zürich, Zurich
  - Universtätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Dellon ES, Collins MH, Bredenoord AJ, Philpott H, Biedermann L, Dulcine M, Nguyen-Cleary T, Su C, Yu J, Tan H, Cataldi F, Wu J, Wang W, Clax P, Woolcott JC, Hirano I. Etrasimod as a treatment for eosinophilic oesophagitis (VOYAGE): a double-blind, placebo-controlled, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2025 Jul;10(7):622-633. doi: 10.1016/S2468-1253(25)00062-7. Epub 2025 May 14. PMID 40381637
- [Derived] Dubinsky MC, Wu J, McDonnell A, Lazin K, Goetsch M, Branquinho D, Modesto I, Armuzzi A. Low Incidence of Macular Edema and Other Ocular Events in the Etrasimod Development Program. J Crohns Colitis. 2025 May 8;19(5):jjae173. doi: 10.1093/ecco-jcc/jjae173. PMID 39575597
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD334-206

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a Double-Blind treatment period (24 weeks) and an Open Label Extension (OLE) period (28 weeks). Participants who were in the placebo group during the Double-Blind treatment period were re-randomized to etrasimod 1 milligram (mg) or etrasimod 2 mg at entry into the Open Label Extension period.
Pre-assignment Details: A total of 262 participants were screened in the study. Out of 262, 154 participants failed screening and 108 participants were randomized and treated.
Groups:
- Experimental: Etrasimod 2 mg: Participants received etrasimod 2 mg tablet orally, once daily for 24 weeks in Double-blind treatment and for 28 weeks in OLE period. Participants were then followed up for safety for up to 4 weeks.
- Experimental: Etrasimod 1 mg: Participants received etrasimod 1 mg tablet orally, once daily for 24 weeks in Double-blind treatment and for 28 weeks in OLE period. Participants were then followed up for safety for up to 4 weeks.
- Placebo Then Etrasimod Any Dose: Participants received etrasimod matching placebo orally, once daily for 24 weeks in Double-blind treatment and re-randomized to receive etrasimod tablet 1 or 2 mg orally, once daily for 28 weeks in OLE period. Participants were then followed up for safety for up to 4 weeks.
- OLE: Placebo Then Etrasimod 2 mg: Participants received etrasimod matching placebo orally, once daily for 24 weeks in Double-blind treatment and re-randomized to receive etrasimod tablet 2 mg orally, once daily for 28 weeks in OLE period. Participants were then followed up for safety for up to 4 weeks.
- OLE: Placebo Then Etrasimod 1 mg: Participants received etrasimod matching placebo orally, once daily for 24 weeks in Double-blind treatment and re-randomized to receive etrasimod tablet 1 mg orally, once daily for 28 weeks in OLE period. Participants were then followed up for safety for up to 4 weeks.
Period: Double-Blind Treatment Period (24 Weeks)
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose | OLE: Placebo Then Etrasimod 2 mg | OLE: Placebo Then Etrasimod 1 mg
Started | 41 | 39 | 28 | 0 | 0
Completed | 30 | 31 | 24 | 0 | 0
Not Completed | 11 | 8 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 5 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 1 | 0 | 0
Period: OLE Period (28 Weeks)
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose | OLE: Placebo Then Etrasimod 2 mg | OLE: Placebo Then Etrasimod 1 mg
Started | 30 | 31 | 0 (Participants received placebo in Double-Blind treatment period were re-randomized into OLE Etrasimod 1 mg and Etrasimod 2 mg groups.) | 12 (Participants received placebo in Double-Blind treatment period were re-randomized into OLE Etrasimod 1 mg and Etrasimod 2 mg groups.) | 12 (Participants received placebo in Double-Blind treatment period were re-randomized into OLE Etrasimod 1 mg and Etrasimod 2 mg groups.)
Completed | 21 | 24 | 0 | 11 | 10
Not Completed | 9 | 7 | 0 | 1 | 2
Not completed — Non-compliance | 1 | 0 | 0 | 0 | 1
Not completed — Other | 1 | 2 | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose | Total
Number analyzed (Participants) | 41 | 39 | 28 | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.6 (9.80) | 39.9 (12.87) | 39.1 (11.65) | 38.1 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 14 | 51
  Male | 21 | 22 | 14 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 0 | 9
  Not Hispanic or Latino | 36 | 34 | 28 | 98
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 39 | 38 | 28 | 105
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Esophageal Peak Eosinophil Count (PEC) at Week 16
Description: Eosinophils was counted in the areas of greatest eosinophil density. Counts were reported as the number of eosinophils/high power field (eos/hpf) and multiple hpfs analyzed until the PEC was clearly identified after taking into account all biopsies from all esophageal levels.
Time Frame: Baseline, Week 16
Population: The Full Analysis Set (FAS) will consist of all randomized participants in the Double-Blind Treatment Period who received at least 1 dose of study treatment. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose
Number analyzed (Participants) | 33 | 35 | 20
Percent change | -58.4 [-86.21 to -26.25] | -39.4 [-71.08 to 78.95] | -21.5 [-57.20 to 55.42]
Statistical Analysis 1: Comparison: Experimental: Etrasimod 2 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.0103, ANCOVA; LS mean difference = -18.54, 95% CI 2-sided [-32.60 to -4.49] — Estimates were from ANCOVA model for rank score of percent change from baseline in esophageal PEC
Statistical Analysis 2: Comparison: Experimental: Etrasimod 1 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.2861, ANCOVA; LS mean difference = -7.53, 95% CI 2-sided [-21.48 to 6.42] — Estimates were from ANCOVA model for rank score of percent change from baseline in esophageal PEC

2. Secondary Outcome: Absolute Change From Baseline in Dysphagia Symptom Questionnaire (DSQ) Score at Week 16
Description: The DSQ was used to measure the frequency and intensity of dysphagia to solid food. DSQ contained 4 questions, all participants used a diary, and responded to Questions 1 (did you eat solid food) and 2 (did food pass slowly or get stuck). If the participant's answer to Question 2 was 'No', the diary ended for that day. If a participant answered 'Yes', he/she advanced to Questions 3 (did you have to do anything to make the food go down or get relief) and 4 (extent to which the participant experienced pain while swallowing). DSQ score = (Sum of points from questions 2+3 in the daily DSQ)×14 days/(Number of diaries reported with non-missing data). DSQ scores can range from 0 to 84, with a higher score indicating worse dysphagia.
Time Frame: Baseline, Week 16
Population: The FAS will consist of all randomized participants in the Double-Blind Treatment Period who received at least 1 dose of study treatment. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose
Number analyzed (Participants) | 32 | 36 | 24
Units on a scale | -17.11 (2.247) | -14.78 (2.166) | -19.49 (2.602)
Statistical Analysis 1: Comparison: Experimental: Etrasimod 2 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.4894, Linear mixed effects model; LS mean difference = 2.38, 95% CI 2-sided [-4.43 to 9.19]
Statistical Analysis 2: Comparison: Experimental: Etrasimod 1 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.1671, Linear mixed effects model; LS mean difference = 4.70, 95% CI 2-sided [-2.00 to 11.41]

3. Secondary Outcome: Absolute Change From Baseline in Esophageal Peak Eosinophil Count (PEC) at Week 16
Description: as for outcome 1
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: eos/hpf
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose
Number analyzed (Participants) | 33 | 35 | 20
eos/hpf | -46.3 (17.46) | -5.7 (16.99) | 8.3 (22.37)
Statistical Analysis 1: Comparison: Experimental: Etrasimod 2 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.0565, ANCOVA; LS mean difference = -54.53, 95% CI 2-sided [-110.59 to 1.54]
Statistical Analysis 2: Comparison: Experimental: Etrasimod 1 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.6193, ANCOVA; LS mean difference = -13.95, 95% CI 2-sided [-69.61 to 41.71]

4. Secondary Outcome: Percentage Of Participants With Esophageal Peak Eosinophil Count (PEC) Less Than (<) 15 Eosinophils/High Power Field (Eos/Hpf) at Week 16
Time Frame: Week 16
Population: The FAS will consist of all randomized participants in the Double-Blind Treatment Period who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose
Number analyzed (Participants) | 41 | 39 | 28
Percentage of participants | 22.0 | 12.8 | 0
Statistical Analysis 1: Comparison: Experimental: Etrasimod 2 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.0007, Mantel Haenszel; Adjusted difference from placebo = 21.90, 95% CI 2-sided [9.23 to 34.57]
Statistical Analysis 2: Comparison: Experimental: Etrasimod 1 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.0121, Mantel Haenszel; Adjusted difference from placebo = 13.85, 95% CI 2-sided [3.03 to 24.66]

5. Secondary Outcome: Percentage of Participants With Esophageal Peak Eosinophil Count (PEC) Less Than or Equal to (<=) 6 Eosinophils/High Power Field (Eos/Hpf) at Week 16
Time Frame: Week 16
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose
Number analyzed (Participants) | 41 | 39 | 28
Percentage of participants | 12.2 | 7.7 | 0
Statistical Analysis 1: Comparison: Experimental: Etrasimod 2 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.0173, Mantel Haenszel; Adjusted difference from placebo = 12.15, 95% CI 2-sided [2.15 to 22.16]
Statistical Analysis 2: Comparison: Experimental: Etrasimod 1 mg vs Placebo Then Etrasimod Any Dose; Test type: Other; p = 0.0590, Mantel Haenszel; Adjusted difference from placebo = 8.37, 95% CI 2-sided [-0.32 to 17.07]

6. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Maximum Severity During 24 Week Double Blind Treatment Period
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AE is defined as an AE that started or worsened in severity on or after the first dose of study treatment. Severity is classified as Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe, Grade 4: Life-Threatening, Grade 5: Death Related to AE.
Time Frame: Baseline, up to Week 24
Population: The safety population included all randomized participants who received at least 1 dose of study treatment during the specified treatment period. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose
Number analyzed (Participants) | 29 | 27 | 21
Participants
  TEAE: Grade 1 | 19 | 15 | 8
  TEAE: Grade 2 | 9 | 12 | 11
  TEAE: Grade 3 | 1 | 0 | 2
  TEAE: Grade 4 | 0 | 0 | 0
  TEAE: Grade 5 | 0 | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Serious TEAEs, TEAEs Leading to Study Treatment Discontinuation, TEAEs Leading to Death and TEAEs of Special Interest During 24 Week Double Blind Treatment Period
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of death); new or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 24 weeks after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to etrasimod was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to Week 24
Population: The safety population included all randomized participants who received at least 1 dose of study treatment during the specified treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose
Number analyzed (Participants) | 41 | 39 | 28
Participants
  Serious TEAEs | 0 | 0 | 0
  TEAEs leading to study treatment discontinuation | 1 | 0 | 1
  TEAEs leading to death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to a maximum of 61 weeks (35 days screening period, 24 weeks of double-blind treatment period, 28 weeks of active extended treatment, and 4 weeks of follow-up period)
Description: Same event may appear as both non-SAE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. All participants who receive any of the study intervention.
Groups:
- OLE: Etrasimod 2 mg: Participants received etrasimod 2 mg tablet orally, once daily for 28 weeks in OLE period. Participants were then followed up for safety for up to 4 weeks.
- OLE: Etrasimod 1 mg: Participants received etrasimod 1 mg tablet orally, once daily for 28 weeks in OLE period. Participants were then followed up for safety for up to 4 weeks.
Arm/Group | Experimental: Etrasimod 2 mg | Experimental: Etrasimod 1 mg | Placebo Then Etrasimod Any Dose | OLE: Etrasimod 2 mg | OLE: Etrasimod 1 mg | OLE: Placebo Then Etrasimod 2 mg | OLE: Placebo Then Etrasimod 1 mg
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39 | 0/28 | 0/30 | 0/31 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39 | 0/28 | 0/30 | 0/31 | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 30/41 | 27/39 | 23/28 | 16/30 | 19/31 | 11/12 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Etrasimod 2 mg (N=41) | Experimental: Etrasimod 1 mg (N=39) | Placebo Then Etrasimod Any Dose (N=28) | OLE: Etrasimod 2 mg (N=30) | OLE: Etrasimod 1 mg (N=31) | OLE: Placebo Then Etrasimod 2 mg (N=12) | OLE: Placebo Then Etrasimod 1 mg (N=12)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Etrasimod 2 mg (N=41) | Experimental: Etrasimod 1 mg (N=39) | Placebo Then Etrasimod Any Dose (N=28) | OLE: Etrasimod 2 mg (N=30) | OLE: Etrasimod 1 mg (N=31) | OLE: Placebo Then Etrasimod 2 mg (N=12) | OLE: Placebo Then Etrasimod 1 mg (N=12)
Nausea (Gastrointestinal disorders) | 6 | 3 | 3 | 2 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 1 | 5 | 0 | 1 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bile acid malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 4 | 4 | 6 | 2 | 5 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0 | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 4 | 1 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 1 | 1 | 1 | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypoglossal nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 0 | 4 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual field defect (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 2 | 1 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acquired oesophageal web (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT04682639/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT04682639/SAP_001.pdf